CLINICAL TRIAL: NCT04269317
Title: A Prospective Study With Blinded Assessment to Evaluate the Safety and Effectiveness of the Tixel C Fractional System in the Treatment of Acne Scars
Brief Title: Clinical Study to Evaluate the Safety and Effectiveness of the Treatment With Tixel C on Acne Scars
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay in opening the study due to COVID-19, and following the sponsor's decision
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0472
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Scars
Keywords: Acne Scars; Post Acne; Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Masking Description: Blinded assessed of the improvement would be done between Last FU images and before first treatment after randomization of the images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tixel C (Experimental): Tixel Treatment, between 3-5 treatment session according to investigator's review of subject response follow by 3 Follow up sessions, 1,3 and 6 month after last treatment visit. Subject would be questioned about pain levvel, subjective dountime assessment and subjective response assessment. Images would be taken before treatment visit and in Follow-Up.
  Interventions: Device: Tixel C

INTERVENTIONS:
Device: Tixel C — Thermo-mechanical technology for fractional treatment of human skin. Dermal heating and coagulative effect that occur during the treatment session provide for dermal remodeling and collagen restructuring that promote acne scar appearance improvement.
  Other Names: Fractional

SUMMARY:
The purpose of this research is to evaluate the safety and effectiveness of the Tixel C device for the treatment of acne scars, for improvement in the appearance of surface texture.

DETAILED DESCRIPTION:
44 participents between two research locations with moderate acne scars will receive 3-5 treatments sessions with the Tixel C device according to investigator's review of subject response. Improvement of acne scarring will ve evaluated at 1 month, 3 months and 6 months post treatment.

Post-treatment response will be evaluated as well as any incidence of side efects throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. The Subjects will have atrophic mild to severe acne scars.
2. Male or female subjects, age 18-65 years old.
3. The subjects will have Fitzpatrick Skin Types I-VI.
4. Willingness and ability to provide written informed consent, including photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup), prior to the study.
5. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
6. Females post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

1. Subjects pregnant or planning to become pregnant, or have given birth less than three months ago or breast feeding.
2. Subjects with significant exposure to ultraviolet light.
3. Use of drugs that may induce hyperpigmentation such as amiodarone, clofazinmine, minocycline or chloroquine.
4. History of facial acne scar treatments with laser, surgical, chemical, light based or radiofrequency facial treatments.
5. Microdermabrasion, or prescription level glycolic acid treatments within three months prior to study participation.
6. Active HSV-1. May be enrolled only after a prophylactic regime has been followed prior to treatment and according to the Investigator's discretion.
7. History of keloid formation.
8. Permanent facial implant over area of treatment.
9. Injectable filler in area to be treated within nine months of investigation.
10. History of collagen vascular disease.
11. Subjects who have an impaired immune system, suffer from immunosuppressive diseases or are actively on immunosuppressive medications.
12. Subjects currently taking or have taken an oral retinoid in the past six months.
13. Subjects currently taking long-term oral steroid treatment
14. Subjects with any skin pathology which can induce bullous lesions, urticaria, or demonstrate a Koebner phenomenon (psoriasis, lichen planus, etc.).
15. History of autoimmune disease.
16. History of any disease that inhibits pain sensation.
17. History of Diabetes I or II.
18. Concurrent therapy that, in the principal investigator's opinion, would interfere with the evaluation of the safety or effectiveness of the study treatment.
19. Subjects who, in the Investigator's opinion, have a history of poor cooperation, non-compliance with medical treatment or unreliability.
20. Enrollment in any active study involving the use of investigational devices or drugs who in the Investigator's opinion would interfere with the evaluation of the current investigative device.
21. Any other contraindication stated in the guidance documents of the treatment device.
22. Any existing skin disease that in the investigator's opinion would interfere with the evaluation of the safety of the study treatment and any other cause per the principal investigator's discretion.
23. Hypertrophic facial acne scarring or other hypertrophic scarring.
24. Failure to acquire adequate baseline and final photography.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Safety Adverse Events report | up to 12 months
  Safety of the investigational device shall be assessed via quantification of the incidence of devicerelated/non-related undesired effects, which shall be documented and reported as an Adverse Event (AE) or as a Serious Adverse Event (SAE). Known undesired effects may be any of the list stated in the previous paragraph of Expected Possible Side Effects, or any other undesired effect, not described in the said list. The incidence of the device related undesired effects should be analyzed considering severity, causal relation to the investigational device and duration, whether it is transient or permanent.
Effectiveness using Goodman and Baron Assessment scale | up to 12 months; Improvement between last follow up and baseline (before first treatment)
  Before starting therapy and at one and six months follow up visits, the subjects shall be photographed using clinical photography equipment. The images shall be evaluated by blinded raters. The evaluation shall be performed by three raters.
  The scores shall be analyzed according to the statistical plan of the study. Scale between 1-4; 1 = Macular, 4= Severe

SECONDARY OUTCOMES:
Performance using Goodman and Baron Assessment scale | up to 12 months; Improvement between last follow up and baseline (before first treatment)
  Live Assessment by a study investigator - In each visit, an investigator or his designee shall examine by observing the subject and photographs will be taken as outlined. Scale between 1-4; 1 = Macular, 4= Severe

CONTACTS AND LOCATIONS:
Overall Officials: Jerome M Garden, MD, Principal Investigator — Physicians Laser and Dermatology Institute
Locations (2):
- Physicians Laser and Dermatology Institute, Chicago, Illinois, United States
- The Lehavit Akerman Main Clinic, Herzliya, Israel